CLINICAL TRIAL: NCT02607098
Title: Understanding Adaptive Challenges Associated With Male-factor Infertility
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00065075
Record Dates: First submitted 2015-11-13; First posted 2015-11-17 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-01

CONDITIONS: Male-factor Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Males diagnosed with male-factor infertility: This study will recruit a convenience sample of 10 men and their partners seeking consultation from a fertility urologist following the detection of male-factor infertility.
- Female partners: This study will recruit a convenience sample of 10 men and their partners seeking consultation from a fertility urologist following the detection of male-factor infertility.

SUMMARY:
The purpose of this study is to understand the experience of men and their partners when diagnosed with male-factor infertility while trying to achieve a pregnancy and the skills they use to adapt to this diagnosis.

ELIGIBILITY:
Inclusion criteria:

Men:

* in a partnered relationship with a female
* have been trying without success to conceive a pregnancy
* have been referred due to suspected or diagnosed male-factor infertility
* have the ability to read and write English

Female Partner:

* 18 to 40 years of age
* ability to read and write English

Exclusion criteria:

* living children, either biological or adoptive
* history of vasectomy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: This study will recruit a convenience sample of 10 men and their partners seeking consultation from a fertility urologist following the detection of male-factor infertility.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2015-11; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Feasibility, as measured by the percentage of eligible subjects agreed to participate | 6 months
Feasibility, as measured by retention percentage | 6 months

SECONDARY OUTCOMES:
Change in level of global infertility stress, as measured by questionnaire | Baseline, 6 months
Change in quality of life, as measured by questionnaire | Baseline, 6 months
Change in level of global infertility stress, as measured by questionnaire | Pre and post significant event, up to 7 months
  The investigators will determine the change in pre and post significant event (when reported, such as new diagnosis, IVF/ICSI, discontinuation of treatment) level of global infertility stress in both the man and his partner.
Change in quality of life, as measured by questionnaire | Pre and post significant event, up to 7 months
  The investigators will determine the change in pre and post significant event (when reported, such as new diagnosis, IVF/ICSI, discontinuation of treatment) level of quality of life in both the man and his partner.
Concordance between men and partners with respect to levels of global infertility stress, as measured by questionnaire | 3 months
Concordance between men and partners with respect to quality of life, as measured by questionnaire | 3 months
Concordance between men and partners with respect to levels of global infertility stress, as measured by questionnaire | 6 months
Concordance between men and partners with respect to quality of life, as measured by questionnaire | 6 months
Feasibility, as measured by percentage of participants who used text messaging to complete their study questionnaires | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Eleanor Stevenson, Ph.D., Principal Investigator — Duke University
Locations (2):
- Duke University Medical Center, Durham, North Carolina, United States
- Newcastle Fertility Centre, Newcastle upon Tyne, England, United Kingdom